CLINICAL TRIAL: NCT03075540
Title: Enhancing At-risk Latina Women's Use of Genetic Counseling for Hereditary Breast and Ovarian Cancer: Using Mental Models to Develop Culturally Targeted Media
Brief Title: Enhancing At-risk Latina Women's Use of Genetic Counseling for Hereditary Breast and Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ADeMendoza
Record Dates: First submitted 2017-02-22; First posted 2017-03-09 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-09

CONDITIONS: Hereditary Breast and Ovarian Cancer
Keywords: Latinas
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome | interventions — Genetic Counseling

STUDY DESIGN:
Intervention Model Description: Single arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YouTube Video (Other): Participants will watch a 15-minute YouTube video. The video will provide information about hereditary breast and ovarian cancer and about the process of genetic counseling and testing.
  Interventions: Behavioral: Genetic Counseling and Testing YouTube Video

INTERVENTIONS:
Behavioral: Genetic Counseling and Testing YouTube Video — Participants (n=40) will watch a 15-minute YouTube video that will describe the genetic counseling and testing process and risk/benefit information in a telenovela style format. Participants will complete pre- and post-assessments. After the session, participants interested in pursuing genetic counseling and testing services will be referred to the patient navigator at their respective sites, who will navigate participants to identified no cost or low cost services

SUMMARY:
Compared to non-Latina Whites, Latinas have a higher prevalence of BRCA1/2 gene mutations but lower use of genetic cancer risk assessments services (GCRA). This study will develop and assess the impact of a novel culturally targeted media intervention to improve psychosocial outcomes and GCRA use in Latinas at-risk of hereditary breast and ovarian cancer. If the intervention is proven to be effective in a future randomized controlled trial, the intervention can be disseminated to clinics and adapted to other ethnic groups.

DETAILED DESCRIPTION:
Breast cancer is the most diagnosed cancer for Latinas and is their leading cause of cancer death. Compared to non-Latina Whites, Latinas are diagnosed younger and with more advanced breast cancer. They also have the second highest prevalence of BRCA1 or BRCA2 gene mutations, that significantly increases their lifetime risk of developing hereditary breast and ovarian cancer (HBOC). The US Preventive Services Task Force recommends referral for genetic cancer risk assessments (genetic counseling and risk assessment as appropriate; GCRA) for women at high risk of carrying a mutation. GCRA informs treatment for survivors and risk management decisions in unaffected women. Latinas have lower GCRA use than Whites.

Explanations for Latinas' suboptimal GCRA participation include environmental (e.g. access) and psychosocial factors (e.g. low knowledge, emotions). There are numerous interventions to promote GCRA use in White populations and the mere handful of interventions that do target Latinas mostly consists of Mexicans or Puerto Ricans. Empirical evidence about successful strategies to improve GCRA uptake is lacking, especially from a growing population of Central/South American immigrants, a group with nuanced different barriers (e.g. social isolation). Our preliminary data suggests that improving access does not necessarily translate into higher GCRA uptake. Our data also highlighted providers' challenges in communicating GCRA risk information given the dearth of genetic materials in Spanish and Spanish-speaking genetic counselors. Media-based tools used to educate Latinas before GCRA are needed. This study will fill these gaps.

To be effective, risk HBOC communication interventions should be anchored within the needs and cultural values of their audience. This is because individuals process risk information in the context of "mental models" - one's intuitive beliefs based on personal experiences and shared cultural knowledge. Mental models influence the interpretation of new information. Often there is incongruence between lay and expert mental risk models that leads to miscommunication and uninformed decision-making. For example, among Latinas, the word "testing" led to the misconception that genetic testing would be repeated akin to other screening tests like mammography. Understanding Latinas' mental models will facilitate targeted risk communication to identify knowledge gaps and reduce misconceptions. Interventions that only address knowledge and/or beliefs may not enhance uptake, as risk information evokes emotional reactions that are often stronger predictors of behaviors than cognitive factors. Anticipated negative emotions to GCRA have been associated with lower uptake. Latinas report ambivalence towards GCRA that may impact their decisions. As most interventions have focused on knowledge and/or access, our study makes a considerable shift in the field by addressing mental models and targeting emotions.

This experienced multidisciplinary team will conduct a risk communication intervention designed to target mental models, emotions, and cultural values. Guided by the Theory of Planned Behavior and Social Cognitive Theory, the investigators will conduct a two-phased mixed methods study. In Phase I the investigators will interview key informants (n=10) and at-risk Latinas (n=20) to describe their mental models and other psychosocial factors. These data will inform the risk-benefit messages that will be evaluated in focus groups (n=20) and used to develop a YouTube-based intervention, which will be delivered via Latina actors and a trusted medical personality. In Phase II the investigators will pilot the intervention on at-risk Latinas (n=40). Participants will complete a baseline survey, watch the 15-minute video, complete a follow-up assessment, and be referred to a patient navigator for resources. The primary outcome is intentions to use GCRA. GCRA uptake will be assessed at 3-months. Specific aims are:

Aim 1. Describe and portray Latinas' GCRA mental models (e.g. risks and benefits perceptions).

Aim 2. Using data from Aim 1, develop the content of the risk-benefit communication messages for at-risk Latinas and incorporate these into a Spanish-language YouTube video.

Aim 3. Evaluate the acceptability and pre- and post-intervention differences on the primary outcome (intentions to use GCRA) and intermediate outcomes (e.g. attitudes). We will also explore post-intervention GCRA uptake as a secondary outcome. H.2.1. The intervention will result in a significant increase in intentions to use GCRA, and in H.2.2. improvements of intermediate outcomes: knowledge, attitudes, self-efficacy, and emotional ambivalence. H.2.3. After the intervention, 30% of Latinas will participate in GCRA by 3-months post-intervention. H.2.4. The majority (≥75%) will be satisfied with the intervention.

This study meets the Healthy People 2020 goals to enhance GCRA in at-risk populations, and the national priorities to increase diversity in genetics research participation and incorporate emotions into cancer research. Findings will inform new strategies for behavioral interventions targeting Latinas and a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Latino/Hispanic, >21 years of age, and are at high risk of carrying a HBOC mutation using personal and family cancer histories based on the National Comprehensive Cancer Network

Exclusion Criteria:

* not having the cognitive ability to provide informed consent

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 88 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Genetic counseling uptake | three months post-intervention
  Participation in genetic counseling services

SECONDARY OUTCOMES:
Intentions Scale | within one hour before the intervention and within one hour post-intervention
  Intentions to use genetic counseling services
Knowledge Scale | within one hour before the intervention and within one hour post-intervention
  Knowledge about hereditary breast and ovarian cancer
Attitudes Scale | within one hour before the intervention and within one hour post-intervention
  Attitudes about participating in genetic counseling services
Self-efficacy Scale | within one hour before the intervention and within one hour post-intervention
  Self-efficacy in participating in genetic counseling services
emotional ambivalence Scale | within one hour before the intervention and within one hour post-intervention
  emotional ambivalence about participating in genetic counseling services

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra H Hurtado de Mendoza, PhD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Capital Breast Care Center, Washington D.C., District of Columbia
  - Nueva Vida, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez-Trillos S, Carrera P, Caballero A, Sheppard VB, Graves KD, Peshkin BN, Schwartz MD, Campos C, Garces N, Mendoza AH. 'How Did That Make You Feel?' Latinas' Use of Genetic Counseling and Testing for Hereditary Cancer Risk After Watching a Culturally Targeted Video and Receiving Patient Navigation. Psychooncology. 2025 Sep;34(9):e70261. doi: 10.1002/pon.70261. PMID 40883500
- [Derived] Gomez-Trillos S, Sheppard VB, Graves KD, Song M, Anderson L, Ostrove N, Lopez K, Campos C, Gonzalez N, Hurtado-de-Mendoza A. Latinas' knowledge of and experiences with genetic cancer risk assessment: Barriers and facilitators. J Genet Couns. 2020 Aug;29(4):505-517. doi: 10.1002/jgc4.1201. Epub 2019 Dec 27. PMID 31883202